CLINICAL TRIAL: NCT01386437
Title: The Natural History and Pathogenesis of Human Fungal Infections
Brief Title: Natural History of Individuals With Immune System Problems That Lead to Fungal Infections
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110187; 11-I-0187
Record Dates: First submitted 2011-06-30; First posted 2011-07-01 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02-02

CONDITIONS: Chronic Mucocutaneous Candidiasis; Invasive Aspergillosis; CARD9; APECED
Keywords: Autoimmune Polyendocrinopathy Candidiasis Ectodermal Dystrophy (APECED); Fungal Infections; Molds; Autoimmune Polyendocrinpathy Syndrome (APS) Type 1; Natural History; Mucocutaneous Fungal Infection; Invasive Fungal Infection
MeSH Terms: conditions — Candidiasis, Chronic Mucocutaneous; Polyendocrinopathies, Autoimmune; Mycoses; Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fungal infections: Patients with or without inherited or acquired abnormalities of immune function manifesting mucocutaneous and/or invasive fungal infections

SUMMARY:
Background:

- The immune system is made up of special cells, tissues, and organs that fight infections. Problems with this system may lead to frequent, severe, or unusual fungal infections. These infections are often difficult to treat. Researchers want to collect blood and tissue samples from people who have unusual, persistent or severe fungal infections or immune problems that increase the risk of these infections.

Objectives:

- To collect medical information and samples for a long-term study of people with immune system problems that lead to fungal infections.

Eligibility:

* People with a history of fungal infections caused by immune system problems.
* Parents, children, and siblings of this group.
* Healthy volunteers not related to the first two groups.

Design:

* This long-term study may last for up to 25 years. Those in the study may need to provide new information about every 6 months. The procedures for each person may vary with the particular diagnosis and the extent of fungal infection. Healthy volunteers may have only one or two visits.
* At the first visit, those in the study will have a full medical history and physical exam. They will also provide blood.
* Research procedures may include the following:
* Saliva, urine or stool testing
* Mouthwash collection for DNA testing
* Collection of cheek cells, nail clippings, or vaginal fluid
* Tests of leftover tissue or body fluid from previous medical procedures
* Skin or oral mucous membrane biopsy
* Collection of white blood cells
* Followup visits will involve a physical exam and updated medical history. Blood, saliva, urine, or nail clipping samples may be taken for ongoing studies. Any additional tests or exams required by the study doctors may also be done.
* Participants may withdraw from the study pool at any time.

DETAILED DESCRIPTION:
This protocol is a natural history study designed to investigate the clinical, microbiologic, genetic and immunologic correlates of primary immune deficiencies and other conditions associated with mucocutaneous and invasive fungal infections (IFIs). The hypothesis is that chronic mucocutaneous mycoses and IFIs are caused by abnormalities in immune function in these patients that can be identified using modern methods in molecular and cell biology and immunology. For inclusion, patients must have a history of or an active mucocutaneous or invasive fungal infection, but may or may not have a defined primary or acquired immunodeficiency state. Patients will undergo evaluations that include history/physical examination and blood, saliva, and possible tissue sampling for genetic and immunological testing. Patient relatives may also be screened for clinical, microbiological, genetic and/or immunological correlates of host defense abnormalities. Healthy volunteers will be enrolled as a source of control blood, saliva, and possible tissue sampling, and for genetic testing.

The aim of this protocol is to use modern methods in molecular and cell biology and immunology to elucidate the immunopathogenesis of fungal disease in humans. A better understanding of primary immunodeficiency and identification of fungal and host risk factors for fungal infection may provide new insights into pathogenesis and identify targets for development of novel therapies. Enrolled subjects may be followed for up to 25 years to undergo additional clinical evaluation and sampling. Follow-up may occur every 6 months or more frequently depending on clinical course, the underlying risk factor(s), and the type of fungal infection. Under some circumstances, standard medical treatment will be provided for a fungal infection or immune deficiency.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients:

Patients with or without inherited or acquired abnormalities of immune function manifesting mucocutaneous and/or invasive fungal infections are eligible for screening and assessment under this protocol. Specifically, patients must meet all the following inclusion criteria in order to participate in this study:

Adults or children (regardless of age, sex, or ethnicity/race) with a known or yet uncharacterized inherited immunodeficiency and a definitively diagnosed mucocutaneous or invasive fungal infection.

OR

Adults or children (regardless of age, sex, or ethnicity/race) with acquired immunodeficiency and a severe, unusual, persistent or treatment-refractory chronic mucocutaneous fungal infection.

OR

Adults or children (regardless of age, sex, or ethnicity/race) with acquired immunodeficiency and a possible, probable or proven invasive fungal infection (European Organization for Research and Treatment of Cancer / Mycoses Study Group criteria).

OR

Adults or children (regardless of age, sex, or ethnicity/race) with a well-documented prior, unusual, severe, persistent, or treatment-refractory mucocutaneous or invasive fungal infection(s), who have clinically recovered from the fungal infection.

OR

Adults or children (regardless of age, sex, or ethnicity/race) with confirmed or suspected autoimmune polyendocrinopathy-candidiasis-ectodermal dystrophy (APECED) who have not yet developed CMC.

Ongoing care by a referring/primary care physician (inside or outside NIH).

Willing to allow storage of blood and tissue samples for future analyses.

Willing to allow genetic testing from blood, body fluids or tissue specimens.

Willing to have HIV testing

Able to provide informed consent or be accompanied by a parent(s)/legal guardian(s) or legally authorized representative (LAR) who is able to provide informed consent.

No children under the age of 2 years will be seen at the Clinical Center, however they will be able to participate via mail-in specimens

Patient Relatives:

Individuals (regardless of age, sex, or ethnicity/race) who are genetically related to the patient (e.g., mother, father, siblings, children) may be recruited to establish the genetic origin of immune defects that may be identified in the study patients at the discretion of the PI. Relatives must meet all the following inclusion criteria in order to participate in this study:

Willing to allow storage of blood and tissue samples for future analyses.

Willing to allow genetic testing from blood, body fluids or tissue specimens.

Willing to have HIV testing

Able to provide informed consent or, if younger than 18, be accompanied by a parent(s)/legal guardian(s) who is able to provide informed consent.

Healthy Volunteers:

Healthy adults regardless of sex, and ethnicity/race between the ages of 18 and 85 years old may be eligible to participate in this study. Healthy volunteers must meet all the following inclusion criteria in order to participate in this study:

Willing to allow storage of blood and tissue samples for future analyses.

Willing to allow genetic testing from blood, body fluids or tissue specimens.

Willing to have HIV testing

Able to provide informed consent

NIH employees are eligible

EXCLUSION CRITERIA:

Patients:

A patient will not be eligible if he/she has any of the following:

Any condition which, in the investigator's opinion, may interfere with the evaluation of a co-existing abnormality of immunity that is the subject of study under this protocol.

Any condition which, in the investigator's opinion, places the patient at undue risk by participating in the study.

Unwillingness to undergo testing or procedures associated with this protocol.

Hemoglobin of < 7 gm/dL. If a patient is enrolled solely to obtain left-over pathology specimens, saliva, a buccal sample, skin swab, vaginal swab, or a stool sample, this exclusion criteria will not apply as there will be no blood withdrawal.

Patient Relatives:

A genetically related relative will not be eligible for this study if he/she has any condition which, in the investigator's opinion, may interfere with the evaluation of an immune system abnormality that is the subject of study under this protocol.

Healthy Volunteers:

A healthy volunteer will not be eligible if he/she has any of the following:

HIV infection.

History of recurrent or severe infections.

History of an underlying malignancy or receipt of cancer chemotherapy within the past 5 years

Receipt of systemic corticosteroids or other systemic immunosuppressants or immunomodulators within the past 30 days

Pregnancy or lactating

History of heart, lung, kidney disease, or bleeding disorders.

Any condition which, in the investigator's opinion, may interfere with the comparison of clinical specimens against those obtained from affected subjects.

Ages: 1 Day to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be drawn from referrals from the NIH Clinical Center staff, physicians at outside medical facilities, the Clinical Center Volunteer Program, and self-referrals. Patients may be evaluated as inpatients, or at the NIAID outpatient clinic depending on the severity of the clinical manifestations of their infection. The patients genetic relatives will be evaluated at the NIAID outpatient clinic. Patients or relatives who meet the inclusion and/or exclusion criteria, but who are not able to travel to the NIH Clinical Center may be enrolled in the study and evaluated for immune and genetic defects using send-in blood samples or clinical specimens (e.g., previously obtained biopsy specimens or saliva). Healthy volunteers must be seen at NIH and will not have the option to mail in samples.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2012-11-05 (Actual)

PRIMARY OUTCOMES:
Immunological mechanisms of fungal susceptibility | 25 years
  Characterize and understand the immunological mechanism(s) by which inherited immunodeficiencies or acquired conditions increase susceptibility to mucocutaneous and invasive fungal infections.

SECONDARY OUTCOMES:
Determine microbiologic test usefullness | 25 years
  Determine the usefulness of various microbiologic tests (e.g., cultures, serology, molecular assays) for diagnosis and follow-up of the course of fungal infections.
Determine immunological profile of mucosal fungal infections | 25 years
  Define the transcriptional profiles and perform proteomic and microbiome analyses of skin, oral and/or vaginal mucosa, and/or other tissues, and body fluids of patients with inherited or acquired conditions predisposing them to fungal infections.

CONTACTS AND LOCATIONS:
Overall Officials: Michail S Lionakis, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ahonen P, Myllarniemi S, Sipila I, Perheentupa J. Clinical variation of autoimmune polyendocrinopathy-candidiasis-ectodermal dystrophy (APECED) in a series of 68 patients. N Engl J Med. 1990 Jun 28;322(26):1829-36. doi: 10.1056/NEJM199006283222601. PMID 2348835
- [Background] Atkinson TP, Schaffer AA, Grimbacher B, Schroeder HW Jr, Woellner C, Zerbe CS, Puck JM. An immune defect causing dominant chronic mucocutaneous candidiasis and thyroid disease maps to chromosome 2p in a single family. Am J Hum Genet. 2001 Oct;69(4):791-803. doi: 10.1086/323611. Epub 2001 Aug 21. PMID 11517424
- [Background] Holland SM, DeLeo FR, Elloumi HZ, Hsu AP, Uzel G, Brodsky N, Freeman AF, Demidowich A, Davis J, Turner ML, Anderson VL, Darnell DN, Welch PA, Kuhns DB, Frucht DM, Malech HL, Gallin JI, Kobayashi SD, Whitney AR, Voyich JM, Musser JM, Woellner C, Schaffer AA, Puck JM, Grimbacher B. STAT3 mutations in the hyper-IgE syndrome. N Engl J Med. 2007 Oct 18;357(16):1608-19. doi: 10.1056/NEJMoa073687. Epub 2007 Sep 19. PMID 17881745
- [Derived] Ferre EMN, Yu Y, Oikonomou V, Hilfanova A, Lee CR, Rosen LB, Burbelo PD, Vazquez SE, Anderson MS, Barocha A, Heller T, Soldatos A, Holland SM, Walkiewicz MA, Lionakis MS. Case report: Discovery of a de novo FAM111B pathogenic variant in a patient with an APECED-like clinical phenotype. Front Immunol. 2023 Feb 17;14:1133387. doi: 10.3389/fimmu.2023.1133387. eCollection 2023. PMID 36875114
- [Derived] Chascsa DM, Ferre EMN, Hadjiyannis Y, Alao H, Natarajan M, Quinones M, Kleiner DE, Simcox TL, Chitsaz E, Rose SR, Hallgren A, Kampe O, Marko J, Ali RO, Auh S, Koh C, Belkaid Y, Lionakis MS, Heller T. APECED-Associated Hepatitis: Clinical, Biochemical, Histological and Treatment Data From a Large, Predominantly American Cohort. Hepatology. 2021 Mar;73(3):1088-1104. doi: 10.1002/hep.31421. PMID 32557834
- [Derived] Burbelo PD, Ferre EMN, Chaturvedi A, Chiorini JA, Alevizos I, Lionakis MS, Warner BM. Profiling Autoantibodies against Salivary Proteins in Sicca Conditions. J Dent Res. 2019 Jul;98(7):772-778. doi: 10.1177/0022034519850564. Epub 2019 May 16. PMID 31095438
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-I-0187.html